CLINICAL TRIAL: NCT02006251
Title: Comparison of Acetabular Shell Position Using Real-Time Instruments vs. Standard Surgical Instruments: A Randomized Clinical Trial
Brief Title: Real-Time Instrument for Acetabular Shell Positioning
Acronym: RTI
Status: Terminated | Type: Interventional
Why Stopped: Discretion of PI
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wael Barsoum, Vice-chairman, Department of Orthopaedic Surgery, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCF 13-940
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Total Hip Arthroplasty
Keywords: Total Hip Arthroplasty; Acetabular positioning; Patient specific instrumentation; Preoperative planning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Standard Total Hip Arthroplasty (Active Comparator): Each surgeon will use their standard methods of pre-operative planning using pre-operative x-rays, and complete the procedure using standard surgical instruments for total hip arthroplasty.
  Interventions: Procedure: Standard Total Hip Arthroplasty
- Real-time Instrumentation (Experimental): Pre-operative planning through 3D software with design of real-time instrument intraoperatively using bone cement and surrogate bone model for placement of a guide pin to be used to aid in bone preparation for insertion of an acetabular cup in total hip arthroplasty
  Interventions: Device: Real-time Instrumentation; Procedure: Standard Total Hip Arthroplasty

INTERVENTIONS:
Device: Real-time Instrumentation — To prepare the acetabulum and place the implants on the day of surgery, surgeons will receive either parts necessary to create the real-time with a surrogate model of the acetabular surface or standard surgical alignment instruments provided by the manufacturer of the implant. For the experimental group, the surgeon will be provided with 3 parts necessary to create the real-time instrument: (1) a patient-specific surrogate bone model with a built-in guide pin trajectory which was planned in the 3D planning software, (2) a non-specific plastic arm available in different sizes, and (3) bone cement. The real-time instrument is created to position a peripheral guide wire on the acetabular rim to serve as a visual aid for reaming and impacting the acetabular shell using standard reaming tools supplied by the manufacturer. Once the acetabular shell is placed, the procedure is performed in the same manner for both groups, using the standard manufacturer instruments.
  Other Names: RTI
  Arms: Real-time Instrumentation
Procedure: Standard Total Hip Arthroplasty — Total hip arthroplasty performed according to standard of care

SUMMARY:
The proposed study is a double-blinded randomized controlled trial comparing Real-time instruments with solely standardized instruments for the placement of the acetabular cup prosthesis used in total hip arthroplasty.

The investigators will enroll 44 patients who have consented to total hip arthroplasty for treatment of hip pathology. This treatment is a standard of care. Patients will receive standard of care pre- and post-operative care and placement of standard of care implants all of which are commercially available and FDA approved for general use for the clinical indications used in these patients. All patients will receive a pre-operative CT scan for surgical planning and comparison with post-operative CT scan. The difference in intervention between the groups will be the creation and use of real-time instrument from the pre-operative planning session. These instruments will be used for placement of an indexing peripheral guide wire to direct acetabular preparation and placement of the shell assisting standard surgical instruments.

The post-operative scan will be performed within two weeks of the surgery for both the treatment and control groups. The investigators will analyze the difference in acetabular shell placement (acetabular version and abduction angle) from the pre-operatively planned CT scan. These differences will be compared between the control and experimental groups.

ELIGIBILITY:
Inclusion Criteria:

Subjects to be included in this protocol will be adult males and females of all races and socioeconomic status meeting the following criteria:

* Primary, unilateral anterior or posterior total hip arthroplasty
* 18 to 85 years old at time of surgery
* Able to get a pre- and post-operative CT scan at the Cleveland Clinic

Exclusion Criteria:

* Significant metal in the joint that results in metal artifact on the pre--operative CT scan, thereby compromising the ability to visualize the acetabulum on the pre-operative simulator.
* Pregnancy
* Incarceration
* Condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Small T, Krebs V, Molloy R, Bryan J, Klika AK, Barsoum WK. Comparison of acetabular shell position using patient specific instruments vs. standard surgical instruments: a randomized clinical trial. J Arthroplasty. 2014 May;29(5):1030-7. doi: 10.1016/j.arth.2013.10.006. Epub 2013 Oct 16. PMID 24231437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Total Hip Arthroplasty | Real-time Instrumentation
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Total Hip Arthroplasty | Real-time Instrumentation | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (15.0) | 59.3 (11.8) | 60.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Planned and Actual Values of Abduction
Description: The overall difference in component placement between standard of care instrumentation and real-time instrumentation will be compared.
Time Frame: Through 2 weeks after surgery.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Standard Total Hip Arthroplasty | Real-time Instrumentation
Number analyzed (Participants) | 10 | 11
degrees | 5.6 (13.0) | 7.5 (9.4)

2. Secondary Outcome: Difference Between Planned and Actual Values of Version
Description: as for outcome 1
Time Frame: Through 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Standard Total Hip Arthroplasty | Real-time Instrumentation
Number analyzed (Participants) | 10 | 11
degrees | 4.1 (7.8) | 0.6 (9.6)

3. Secondary Outcome: Difference in the Time for Acetabular Preparation and Shell Placement Between the Two Groups
Description: Difference in the time for acetabular preparation and shell placement between the two groups were not collected
Time Frame: Intraoperatively (during surgery)
Population: These data were not collected
Arm/Group | Standard Total Hip Arthroplasty | Real-time Instrumentation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard Total Hip Arthroplasty | Real-time Instrumentation
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Total Hip Arthroplasty (N=10) | Real-time Instrumentation (N=11)
Fall followed by dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient fell and dislocated the hip prosthesis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes